CLINICAL TRIAL: NCT01448980
Title: The Efficacy of Thai Traditional Massage in Decreasing Spasticity for Elderly With Stroke
Brief Title: Efficacy of Massage in Stroke Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Vilai Kuptniratsaikul, Rehabilitation Medicine Department, Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si205/2011
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Stroke; Sequelae
Keywords: massage; stroke spasticity
MeSH Terms: conditions — Stroke | interventions — Medicine, Thai Traditional; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical therapy (Active Comparator): The control group will receive physical therapy 2 time per week for 6 weeks
  Interventions: Procedure: Physical therapy program
- Thai Traditional Massage (Experimental): The experimental group will receive Thai traditional massage program 2 times per week for 6 weeks.
  Interventions: Procedure: Thai Traditional Massage (TTM)

INTERVENTIONS:
Procedure: Thai Traditional Massage (TTM) — Thai Traditional Massage will receive massage 2 time per week for 6 weeks
  Other Names: Thai Traditional Massage
  Arms: Thai Traditional Massage
Procedure: Physical therapy program — Physical therapy program 2 times per week for 6 weeks.
  Other Names: Physical therapy
  Arms: Physical therapy

SUMMARY:
Stroke is one of the common diseases in the elderly. It is the third ranking cause of death and affects health care system in our country. One of the most important consequences of stroke is spasticity. Some stroke patients suffered from severe spasticity or hypersensitive reflex to stimuli. It can cause contracture, limit self care function, transfer or ambulation. Most of stroke patients have to depend on their relatives or families.

DETAILED DESCRIPTION:
Thai traditional massage is one of the popular alternative medicine in Thailand. Lots of stroke patients who suffered from spasticity sought treatment. To the investigators knowledge, there is no study concerning efficacy of massage in decreasing spasticity for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Stroke with onset of >=6 months
* Age >=50 years
* Spasticity grade of knee flexor or elbow flexor was 2-3 classified by Modified Ashworth scale (MAS)
* Ability to follow command and communicable

Exclusion Criteria:

* Having contraindications for massage including fever > 38 degree, uncontrolled blood pressure, bleeding tendency, on anticoagulant drug, having ulcer or healing fracture of limbs, contamination skin disease, severe osteoporosis
* Serious contact diseases, for example AIDS, TB
* History of malignancy
* Fixed joint contracture at elbow or knee of paralyzed limb
* History of botulinum toxin injection or Phenol/Alcohol nerve block within 3 months
* Previous history of TTM
* Severe dementia or uncontrolled psychiatric problems

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth scale (MAS) | 6 weeks
  The massage will be considered success if MAS decreased at least 1 level after treatment.

SECONDARY OUTCOMES:
Modified Barthel index (BI) | 6 weeks
  Massage will be considered success if BI score increases after treatment.
Hospital anxiety depression score (HADS) | 6 weeks
  Massage will be considered success if HADS decreases after treatment.
Thai Pictorial Quality of Life questionnaire | 6 weeks
  Massage will be considered if Thai pictorial QoL score increases after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Vilai Kuptniratsaikul, MD, Principal Investigator — Rehabilitation Medicine Department, Siriraj Hospital, Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Thanakiatpinyo T, Suwannatrai S, Suwannatrai U, Khumkaew P, Wiwattamongkol D, Vannabhum M, Pianmanakit S, Kuptniratsaikul V. The efficacy of traditional Thai massage in decreasing spasticity in elderly stroke patients. Clin Interv Aging. 2014 Aug 11;9:1311-9. doi: 10.2147/CIA.S66416. eCollection 2014. PMID 25143717